CLINICAL TRIAL: NCT00320476
Title: Velcade®, Thalidomide, Dexamethasone (VTD) Induction Therapy Followed By Melphalan, Prednisone, Thalidomide (MPT) Maintenance As a First Line Treatment For The Patients With Multiple Myeloma Who Are Non-Transplant Candidates
Brief Title: VTD Followed By MPT Maintenance As a First Line Treatment For The Patients With MM Who Are Non-Transplant Candidates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korean Multiple Myeloma Working Party (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Lee M.D., korean Multiple Myeloma Working Party
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMM52; 26866138MMY2027
Record Dates: First submitted 2006-04-27; First posted 2006-05-03 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2006-04

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Velcade

SUMMARY:
Multiple Myeloma is a incurable disease. Recently developed targeted therapy gave new hope for the patients with multiple myeloma. Velcade in combination with other agents are currently in trials for the newly diagnosed patient, we designed sequential treatment with VTD and MPT for the patients who are not transplant candidates. This would be expected to result in maximal tumor control, and thus, in maximal survival benefit, equivalent to high dose therapy with autologous transplantation in younger population

DETAILED DESCRIPTION:
The two effective and non-cross resistant regimens, VTD and MPT, will be applied sequentially to the patients with multiple myeloma who are not transplant candidates. This would be expected to result in maximal tumor control, and thus, in maximal survival benefit, equivalent to high dose therapy with autologous transplantation in younger population

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with overt multiple myeloma who are not candidates for HDT/SCT because of old age (> 65) or presence of comorbid conditions likely to have a negative impact on tolerability of HDT/SCT. Sponsors review this conditions and approval is required.
* Presence of measurable disease : serum M-protein > 1g/dL or urine M- protein > 400mg/day
* Performance status £ ECOG 2
* Expected survival ³ 6 months
* Pretreatment clinical laboratory values meeting the following criteria within 14 days before enrollment platelet ≥ 100 x 109/L hemoglobin ≥ 8 g/dL (≥ 4.96 mol/L) Prior RBC transfusion or recombinant human erythropoietin use is allowed) absolute neutrophil count (ANC) ≥ 1.0 x 109/L aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal total bilirubin ≤ 1.5 times the upper limit of normal serum creatinine ≤ 3mg/dL corrected serum calcium <14 mg/dL (<3.5 mmol/L)
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Smoldering or indolent myeloma
* History of allergic reaction attributable to compounds containing boron or mannitol
* Known hypersensitivity to thalidomide or dexamethasone
* Peripheral neuropathy or neuropathic pain Grade 2 or higher as defined by NCI CTCAE version 3
* Uncontrolled or severe cardiovascular disease, including MI within 6 months of enrolment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, or cardiac amyloidosis, cardiac ejection fraction <0.5 : Severe conduction disorder : Hypotension (sitting systolic BP ≤ 100 mmHg and/or sitting diastolic BP ≤ 60 mmHg
* Sepsis
* Pregnancy or breastfeeding
* Uncontrolled Diabetes Mellitus
* Recurrent DVT or pulmonary embolism
* Active ulcers detected by gastroscopy
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Receipt of extensive radiation therapy within 4 weeks

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-04; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response rate of VTD induction Therapy | 2008-02-01

SECONDARY OUTCOMES:
Response rate of VTD/MPT maintenance therapy | 2008-02-01
Progression free survival Overall survival of VTD/MPT | 2008-02-01
To evaluate toxicities of VTD/MPT | 2008-02-01

CONTACTS AND LOCATIONS:
Overall Officials: Jae Hoon Lee, M.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Gachon University Gil Hospital, Inchon, South Korea

REFERENCES:
- [Derived] Eom HS, Kim YK, Chung JS, Kim K, Kim HJ, Kim HY, Jin JY, Do YR, Oh SJ, Suh C, Seong CM, Kim CS, Lee DS, Lee JH. Bortezomib, thalidomide, dexamethasone induction therapy followed by melphalan, prednisolone, thalidomide consolidation therapy as a first line of treatment for patients with multiple myeloma who are non-transplant candidates: results of the Korean Multiple Myeloma Working Party (KMMWP). Ann Hematol. 2010 May;89(5):489-97. doi: 10.1007/s00277-009-0871-y. Epub 2009 Dec 10. PMID 20012045